CLINICAL TRIAL: NCT04452188
Title: Targeting Normoxia in Neonates With Cyanotic Congenital Heart Disease in the Intra-operative and Immediate Post-operative Period (T-NOX)
Brief Title: Targeting Normoxia in Neonates With Cyanotic Congenital Heart Disease in the Intra-operative and Immediate Post-operative Period
Acronym: T-NOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nathaniel Sznycer-Taub, Assistant Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00175086; 5UL1TR002240-05 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Hypoplastic Left Heart Syndrome; Total Anomalous Pulmonary Venous Return; Truncus Arteriosus; Pulmonary Atresia With Ventricular Septal Defect; Transposition of the Great Arteries; Double Outlet Right Ventricle, Subpulmonary VSD; Tetralogy of Fallot; Double Outlet Right Ventricle With Subaortic Ventricular Septal Defect and Pulmonary Stenosis; Cardiopulmonary Bypass
Keywords: Open heart surgery
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Scimitar Syndrome; Truncus Arteriosus, Persistent; Pulmonary Atresia With Ventricular Septal Defect; Transposition of Great Vessels; Double Outlet Right Ventricle; Tetralogy of Fallot; Pulmonary Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normoxia (Experimental): On bypass, goal PaO2 on cardiopulmonary bypass of 60-100 mm Hg using lower fraction of inspired oxygen (FiO2) (blended sweep gas) via oxygenator
  Post-bypass, goal of PaO2 <100 mm Hg by anesthesia and in ICU via oxygen titration via mechanical ventilator for 24 hours post-op.
  Interventions: Other: Normoxia (with controlled re-oxygenation)
- Standard of care (Active Comparator): Frequent blood gases will be checked per protocol on bypass and correlated with the blood parameter monitoring system to maintain a PaO2 of 200-300 per standard practice
  Interventions: Other: Standard of care ventilation

INTERVENTIONS:
Other: Normoxia (with controlled re-oxygenation) — Participants will receive lower levels of oxygen during surgery and after surgery on the ventilator.
  As cardiopulmonary bypass is being weaned, anesthesia will initiate mechanical ventilation with an FiO2 of 50% or less (unless clinically necessary) to achieve oxygen saturation and PaO2 goals that fit within the expected range for the participant's physiology:
  1. Single ventricle patients (PaO2:35-45 and oxygen saturation 75%-85%)
  2. Two ventricle patients (PaO2: 60-100 and oxygen saturation >92%)
  Arms: Normoxia
Other: Standard of care ventilation — As cardiopulmonary bypass is being weaned, anesthesia will initiate mechanical ventilation per standard protocols. Ventilation will be continued in the ICU and adjusted per standard goals per the intensivist.
  Arms: Standard of care

SUMMARY:
This clinical trial is studying the use of different levels of oxygen exposure during and after cardiopulmonary bypass in eligible infants to learn about its safety during heart surgery.

In addition to having the various doses of oxygen, participants will also have blood samples, ultrasounds of the head, and brain wave patterns monitored.

The hypotheses of this trial are:

* that there will be no difference with regards to adverse events between the infants in the normoxia group compared to the infants in the standard of care group
* there will be a significant difference in the measured partial pressure of oxygen (PaO2) values between the two treatment groups.
* the use of normoxia during cardiopulmonary bypass and in the immediate post-operative period will result in clinically significant decrease in oxidative stress as measured by thiobarbituric acid reactive substances (TBARS) after cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Age less than 30 days of age at time of surgery with need for cardiopulmonary bypass with cardioplegic arrest (with or without deep hypothermic circulatory arrest)
* Diagnosis with cyanosis at baseline (pre-operative PaO2 of less than 50mmHG) due to:

  * Complete admixture lesion (example: hypoplastic left heart syndrome, total anomalous pulmonary venous return, truncus arteriosus, pulmonary atresia with VSD)
  * Transposition physiology (example: D-Transposition of the great arteries or Double outlet right ventricle with subpulmonary VSD)
  * Right-to-left shunt (example: Tetralogy of Fallot, double outlet right ventricle with subaortic VSD and pulmonary stenosis)

Exclusion Criteria:

* Corrected gestation at time of surgery less than 37 weeks
* Prior cardiac arrest
* Current or prior history of extracorporeal membrane oxygenation (ECMO) support
* Current or prior history of needing renal replacement therapy with dialysis
* Prior cardiac surgery requiring cardiopulmonary bypass
* Diagnosis of Ebstein's Anomaly
* Known genetic syndrome other than Trisomy 21 or DiGeorge Syndrome

Max Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Sznycer-Taub, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Normoxia: On bypass, goal PaO2 on cardiopulmonary bypass of 60-100 mm Hg using lower fraction of inspired oxygen (FiO2) (blended sweep gas) via oxygenator
  Post-bypass, goal of PaO2 <100 mm Hg by anesthesia and in ICU via oxygen titration via mechanical ventilator for 24 hours post-op.
  Normoxia (with controlled re-oxygenation): Participants will receive lower levels of oxygen during surgery and after surgery on the ventilator.
  As cardiopulmonary bypass is being weaned, anesthesia will initiate mechanical ventilation with an FiO2 of 50% or less (unless clinically necessary) to achieve oxygen saturation and PaO2 goals that fit within the expected range for the patient's physiology:
  1. Single ventricle patients (PaO2:35-45 and oxygen saturation 75%-85%)
  2. Two ventricle patients (PaO2: 60-100 and oxygen saturation >92%)
Period: Overall Study
Arm/Group | Normoxia | Standard of Care
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants assigned to the Normoxia arm of the study were to have a goal PaO2 of 60-100mmHg during cardiopulmonary bypass and 24 hours post-operation. Of the 15 participants, 1 was taken off protocol due to a cardiac arrest during surgery. Once the participant was stabilized, the protocol was resumed. This protocol deviation was extensively reviewed by the study's DSMB. The decision was made to include the participant's data in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normoxia | Standard of Care | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 5 [4 to 9] | 5 [3 to 8] | 5 [4 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Systemic Oxidative Stress Based on Thiobarbituric Acid Reactive Substances (TBARS)
Description: Oxidative stress (OS) reflects an imbalance between the production and accumulation of reactive oxygen species. Oxidation of lipids leads to the generation of lipid peroxides which can be detected as Thiobarbituric acid reactive substances (TBARS). Thus, levels of serum TBARS were assessed in participants as indicators of OS.
  TBARS levels were assessed at three separate time points in the first 24 hours after surgery (2, 6, and 24 hours). Each participant's post-operative (PO) samples were normalized to their baseline pre-operative sample and described as a fold-of-change from baseline. The fold-of-change describes how much a quantity changes between an original and a subsequent measurement and is calculated as TBARS level at each PO time point / TBARS at baseline.
  The mean values of the fold of change from baseline between the two groups at each PO time-point were compared.
Time Frame: Up to 24 hours following surgery
Measure: Mean (Standard Deviation); unit: Fold Change from Baseline
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Fold Change from Baseline
  2 hours Post-Op (PO) | 1.21 (0.26) | 1.93 (0.63)
  6 hours PO | 1.09 (0.25) | 1.77 (0.7)
  24 hours PO | 0.96 (0.16) | 1.41 (0.29)
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Each participant's post-operative samples were normalized to their baseline sample and described as a fold-of-change from baseline; Test type: Equivalence — Prior studies suggest a 25-50% reduction in oxidative stress in normoxia relative to supra-physiologic oxygen. A 20% difference was considered clinically meaningful, and a sample size of 42 total participants was anticipated to achieve at least 80% power with a two-sided 5% significance level. However, an interim analysis recommended by the DSMB after enrollment of 29 patients revealed a significant difference in the primary outcome between the groups, and enrollment was thus stopped; p < 0.01, t-test, 2 sided — To provide a more conservative estimate of significance, the Hochberg sequential procedure was used for adjustment of multiple comparisons in the serum biomarker data including the primary outcome

2. Primary Outcome: Rate of Observed Adverse Events Between the Two Groups
Description: The count of each of the adverse events within 30 days after the index cardiac surgery, listed here: mortality, cardiac arrest, need for mechanical circulatory support, seizures (clinical or subclinical based on EEG), and need for dialysis is presented below.
Time Frame: 30 days after surgery
Population: A patient can have more than one of the outcomes listed.
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants
  Need for Mechanical Circulatory Support | 1 | 3
  Cardiac Arrest | 1 | 2
  Mortality | 1 | 1
  Need for dialysis | 1 | 1
  Seizure | 2 | 1

3. Primary Outcome: Post-operative Length of Stay
Description: Calculated as number of days in the hospital after surgery.
Time Frame: 30 days after surgery
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Days | 15 [9 to 21] | 15.5 [10 to 21]
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Wilcoxon rank sum test was used to compare the post-operative length of stay between the two groups; Test type: Other; p = 0.66, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Days Alive and Out of the Intensive Care Unit (ICU) at 30 Days After Surgery
Description: This composite measure reflects the number of days alive and not admitted to the ICU. Non-survivors at day 30 were considered to have no ICU-free days.
Time Frame: 30 days after surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
days | 22 [19 to 26] | 22.5 [9 to 26]
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Wilcoxon rank sum test was used to compare the days alive and out of ICU at 30 days since surgery between the two groups; Test type: Other; p = 0.66, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Composite Outcome of Major Adverse Events
Description: The composite endpoint assessed in this study combines in-hospital mortality, cardiac arrest, ECMO, seizures, and dialysis and reflects the number of participants affected by one or more of these outcomes.
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants | 3 | 3
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Test type: Other; p = 1.00, Fisher Exact

6. Primary Outcome: Global Rank Score
Description: Per NCT03229538, a composite mortality, major morbidity and length of stay global rank endpoint with endpoints ranked according to severity. For this endpoint, each randomized patient will be assigned a rank based upon their most-severe outcome. Rank of 91= Post-operative length of stay > 90 days, 92= Post-op cardiac arrest, multi-system organ failure, renal failure with temporary dialysis, or prolonged ventilator support, 93= Reoperation for bleeding, unplanned delayed sternal closure, or post-op unplanned interventional cardiac catheterization, 94= Post-operative mechanical circulatory support or unplanned cardiac reoperation (exclusive of reoperation for bleeding), 95= Renal failure with permanent dialysis, neurologic deficit persistent at discharge, or respiratory failure requiring tracheostomy; 96= Heart transplant (during hospitalization); 97= Operative mortality. Ranks 1 through 90 correspond to the post-operative length of stay in days. A lower score means a better outcome.
Time Frame: 30 days after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Normoxia: On bypass, goal PaO2 on cardiopulmonary bypass of 60-100 mm Hg using lower fraction of inspired oxygen (FiO2) (blended sweep gas) via oxygenator
  Post-bypass, goal of PaO2 <100 mm Hg by anesthesia and in ICU via oxygen titration via mechanical ventilator for 24 hours post-op.
  Normoxia (with controlled re-oxygenation): Participants will receive lower levels of oxygen during surgery and after surgery on the ventilator.
  As cardiopulmonary bypass is being weaned, anesthesia will initiate mechanical ventilation with an FiO2 of 50% or less (unless clinically necessary) to achieve oxygen saturation and PaO2 goals that fit within the expected range for the participant's physiology:
  1. Single ventricle patients (PaO2:35-45 and oxygen saturation 75%-85%)
  2. Two ventricle patients (PaO2: 60-100 and oxygen saturation >92%)
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
score on a scale | 15 [10 to 20] | 17 [10 to 80]
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Test type: Other; p = 0.49, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Systemic Oxidative Stress Based on Protein Carbonyl Levels After Surgery
Description: Protein carbonyls are generated upon oxidation of proteins and are a marker of oxidative stress. Serum protein carbonyl contents were assessed at three separate time points in the first 24 hours after surgery (2, 6, and 24 hours). Each participant's post-operative (PO) samples were normalized to their baseline sample and described as a fold-of-change from baseline. The mean values of the fold of change from baseline between the two groups at each PO time-point were compared. The fold-of-change describes how much a quantity changes between an original and a subsequent measurement and is calculated as Protein Carbonyl level at each PO time point / Protein Carbonyl at baseline.
Time Frame: Up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: Fold Change from Baseline
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Fold Change from Baseline
  2 hours PO | 0.87 (0.25) | 1.3 (0.35)
  6 hours PO | 0.95 (0.3) | 1.6 (0.47)
  24 hours PO | 0.86 (0.2) | 1.7 (0.76)
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Test type: Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

8. Other Pre Specified Outcome: Systemic Oxidative Stress Based on Total Antioxidant Capacity (TAC)
Description: TAC assays measure serum antioxidants in biological samples. Therefore, lower values reflect depletion of antioxidants in the setting of oxidative stress. Serum TAC was assessed at three separate time points in the first 24 hours after surgery (2, 6, and 24 hours). Each participant's post-operative (PO) samples were normalized to their baseline sample and described as a fold-of-change from baseline. The mean values of the fold of change from baseline between the two groups at each PO time-point were compared. The fold-of-change describes how much a quantity changes between an original and a subsequent measurement and is calculated as TAC level at each PO time point / TAC at baseline.
Time Frame: Up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: Fold Change from Baseline
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Fold Change from Baseline
  2 hours PO | 1.3 (0.38) | 0.79 (0.27)
  6 hours PO | 1.4 (0.42) | 0.87 (0.33)
  24 hours PO | 1.4 (0.46) | 0.88 (0.23)
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Test type: Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

9. Other Pre Specified Outcome: Systemic Oxidative Stress Based on 8-Isoprostane Levels After Surgery
Description: 8-isoprostane is a stable oxidative stress marker formed by non-enzymatic perioxidation of lipids. Serum levels of 8-isoprostane were assessed at three separate time points in the first 24 hours after surgery (2, 6, and 24 hours). Each participant's post-operative (PO) samples were normalized to their baseline sample and described as a fold-of-change from baseline. The mean values of the fold of change from baseline between the two groups at each PO time-point were compared. The fold-of-change describes how much a quantity changes between an original and a subsequent measurement and is calculated as 8-isoprostane level at each PO time point / 8-isoprostane at baseline.
Time Frame: Up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: Fold Change from Baseline
Arm/Group | Normoxia | Standard of Care
Number analyzed (Participants) | 15 | 14
Fold Change from Baseline
  2 hour post-operative (PO) | 0.52 (0.41) | 0.89 (0.52)
  6 hours PO | 0.60 (0.50) | 1.0 (0.69)
  24 hours PO | 0.44 (0.37) | 1.1 (1.4)
Statistical Analysis 1: Comparison: Normoxia vs Standard of Care; Test type: Other; p < 0.1, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From time of surgery to 30 days post-operation
Description: Because all of these neonates had just undergone surgery and have many kinds of complications, the IRB approved our collection of a limited set of adverse events. All collected adverse events are shown here.
Arm/Group | Normoxia | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/14
Serious Adverse Events (participants affected / at risk) | 3/15 | 3/14
Other Adverse Events (participants affected / at risk) | 7/15 | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normoxia (N=15) | Standard of Care (N=14)
Cardiac arrest requiring CPR and medications (Cardiac disorders) | 1 | 2
Cardiopulmonary insufficiency requiring ECMO (Cardiac disorders) | 1 | 3
Seizures (Nervous system disorders) | 2 | 1
Need for dialysis (Renal and urinary disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normoxia (N=15) | Standard of Care (N=14)
Post-op Arrhythmias requiring treatment (Cardiac disorders) | 7 | 3
Post-up Stroke (Nervous system disorders) | 0 | 1
Post-op Hemorrhage (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT04452188/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT04452188/ICF_000.pdf